CLINICAL TRIAL: NCT01545583
Title: Study of the Safety, Tolerability and Pharmacokinetics of LY3016859 After Single Intravenous and Subcutaneous Dosing in Healthy Volunteers
Brief Title: A Study of LY3016859 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14352; 2011-005596-17 (EudraCT Number); I5V-MC-TGAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-03-01; First posted 2012-03-07 (Estimated); Results first posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2017-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- Placebo intravenous (Placebo Comparator): Placebo administered once intravenously
  Interventions: Drug: Placebo intravenous
- 0.1 milligram (mg) LY3016859 intravenous (Experimental): 0.1 mg LY3016859 administered once intravenously
  Interventions: Drug: LY3016859 intravenous
- 1 mg LY3016859 intravenous (Experimental): 1 mg LY3016859 administered once intravenously
  Interventions: Drug: LY3016859 intravenous
- 10 mg LY3016859 intravenous (Experimental): 10 mg LY3016859 administered once intravenously
  Interventions: Drug: LY3016859 intravenous
- 50 mg LY3016859 intravenous (Experimental): 50 mg LY3016859 administered once intravenously
  Interventions: Drug: LY3016859 intravenous
- 250 mg LY3016859 intravenous (Experimental): 250 mg LY3016859 administered once intravenously
  Interventions: Drug: LY3016859 intravenous
- 750 mg LY3016859 intravenous (Experimental): 750 mg LY3016859 administered once intravenously
  Interventions: Drug: LY3016859 intravenous
- Placebo subcutaneous (Placebo Comparator): Placebo administered once subcutaneously
  Interventions: Drug: Placebo subcutaneous
- 50 mg LY3016859 subcutaneous (Experimental): 50 mg LY3016859 administered once subcutaneously
  Interventions: Drug: LY3016859 subcutaneous

INTERVENTIONS:
Drug: LY3016859 intravenous — Administered intravenously
  Arms: 0.1 milligram (mg) LY3016859 intravenous; 1 mg LY3016859 intravenous; 10 mg LY3016859 intravenous; 250 mg LY3016859 intravenous; 50 mg LY3016859 intravenous; 750 mg LY3016859 intravenous
Drug: Placebo intravenous — Administered intravenously
  Arms: Placebo intravenous
Drug: LY3016859 subcutaneous — Administered subcutaneously
  Arms: 50 mg LY3016859 subcutaneous
Drug: Placebo subcutaneous — Administered subcutaneously
  Arms: Placebo subcutaneous

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of LY3016859 administered as single doses, and to determine how long LY3016859 remains in the body

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women of non-childbearing potential as determined by medical history and physical examination (PE), and:

  * Men agree to use 2 medically accepted methods of contraception with all sexual partners during the study and for 90 days after the final dose
  * Women are not of child-bearing potential due to surgical sterilization (at least 6 weeks after surgical bilateral oophorectomy with or without hysterectomy or at least 6 weeks after tubal ligation) confirmed by medical history, or post-menopause. Post-menopausal status will be defined as a woman 45 years of age or older with either 12 months of spontaneous amenorrhea, or 6-12 months of spontaneous amenorrhea combined with follicle stimulating hormone (FSH) greater than (>) 40 international units per liter (IU/L)
* Are reliable and are willing to make themselves available for the duration of the study, and are willing to follow site specific study procedures
* Must weigh greater than or equal to (≥) 50 kilograms (kg) at time of screening and dosing
* Have clinical laboratory test results within normal reference range for the investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Have venous access sufficient to allow blood sampling as per the protocol
* Must be a non-smoker

Exclusion Criteria:

* Are currently enrolled in, or have discontinued within the last 60 days from a clinical trial involving an investigational drug that has not received regulatory approval for any indication, or have received treatment with biologic agents (such as monoclonal antibodies) within 3 months or 5 half-lives of the administered drug (whichever is longer) prior to dosing
* Have previously completed or withdrawn from this study or any other study investigating LY3016859, and have previously received the investigational product
* Have a history or presence of medical illness including but not limited to any cardiovascular, hepatic, respiratory, hematological, endocrine, psychiatric or neurological disease, or any clinically significant laboratory abnormality, that in the judgment of the investigator indicates a medical problem that would preclude study participation
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study or have:

  * Confirmed corrected QT interval using Fridericia's formula (QTcF) > 450 milliseconds (msec) for men and > 470 msec for women
  * Bundle branch blocks or other conduction abnormalities other than mild first-degree atrio-ventricular block
  * Irregular rhythms other than sinus arrhythmia or occasional, rare supraventricular ectopic beats
  * History of unexplained syncope
  * Family history of unexplained sudden death or sudden death due to long QT syndrome
  * T-wave configurations are not of sufficient quality for assessing QT interval, as determined by the investigator
* Show evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies, hepatitis C and/or positive hepatitis C antibody, or Hepatitis B and/or positive Hepatitis B surface antigen
* Show use of any medication with potential to mask allergic response for example (e.g.) antihistamines, systemic glucocorticoids or antipyretic agents) within 3 days of dosing (Note: Acetaminophen or nonsteroidal analgesics for headache may be allowed as needed in the Investigator's judgment. The following medications are also specifically allowed in this study: vitamins at normal replacement doses, hormone replacement therapies e.g. estrogen, thyroid hormone), topical medications with limited systemic effects (e.g. eye drops, skin creams, vaginal antifungals, hemorrhoid preparations, etcetera (etc.), stable preventive therapies for hyperlipidemia and gastric acidity disorders)
* Have donated blood of more than 500 milliliters (mL) within the last month.
* Have an average weekly alcohol intake that exceeds 21 units per week or are unwilling to stop alcohol within 48 hours of entry into study and for the duration of the study [1 unit = 12 ounces (oz) or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits]
* Have an abnormal blood pressure (sitting) defined as diastolic blood pressure (DBP) > 95 or less than (<) 50 millimeters of mercury (mmHg) and/or systolic blood pressure (SBP) > 150 or < 90 mmHg confirmed by at least 1 repeat measurement
* Have evidence of regular use of known drugs of abuse or show positive findings for such use on urinary drug screening
* Will donate blood or participate in another clinical trial within 3 months or 5 half-lives of study drug (whichever is longer) of receiving the last study drug administration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern Time (UTC/GMT- 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo IV: Placebo administered once intravenously (IV).
- Placebo SC: Placebo administered once subcutaneously (SC).
- 0.1 mg LY3016859 IV: 0.1 milligram (mg) LY3016859 administered once intravenously.
- 1 mg LY3016859 IV: 1 mg LY3016859 administered once intravenously.
- 10 mg LY3016859 IV: 10 mg LY3016859 administered once intravenously.
- 50 mg LY3016859 IV: 50 mg LY3016859 administered once intravenously.
- 250 mg LY3016859 IV: 250 mg LY3016859 administered once intravenously.
- 750 mg LY3016859 IV: 750 mg LY3016859 administered once intravenously.
- 50 mg LY3016859 SC: 50 mg LY3016859 administered once subcutaneously.
Period: Overall Study
Arm/Group | Placebo IV | Placebo SC | 0.1 mg LY3016859 IV | 1 mg LY3016859 IV | 10 mg LY3016859 IV | 50 mg LY3016859 IV | 250 mg LY3016859 IV | 750 mg LY3016859 IV | 50 mg LY3016859 SC
Started | 12 | 2 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Received at Least 1 Dose of Study Drug | 12 | 2 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 12 | 2 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo IV | Placebo SC | 0.1 mg LY3016859 IV | 1 mg LY3016859 IV | 10 mg LY3016859 IV | 50 mg LY3016859 IV | 250 mg LY3016859 IV | 750 mg LY3016859 IV | 50 mg LY3016859 SC | Total
Number analyzed (Participants) | 12 | 2 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.8 (9.19) | 27.0 (11.31) | 29.7 (8.48) | 36.5 (9.71) | 30.2 (8.59) | 43.2 (17.42) | 41.3 (17.25) | 47.0 (14.68) | 33.0 (11.68) | 35.3 (13.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 5
  Male | 11 | 2 | 6 | 5 | 6 | 4 | 5 | 6 | 6 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 12 | 2 | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 54
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 0 | 0 | 2 | 1 | 2 | 0 | 1 | 1 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 7
  White | 3 | 1 | 5 | 4 | 2 | 3 | 5 | 3 | 4 | 30
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 6
Region of Enrollment [Number; unit: participants]
  United Kingdom | 12 | 2 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 56

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Drug-Related Treatment-Emergent Adverse Events (TEAEs) or Any Serious AEs (SAE)
Description: Drug-related TEAEs are any untoward medical occurrence that either occurs or worsens at any time after treatment baseline, and in the opinion of the investigators is possibly related to study drug. A summary of SAEs and other nonserious AEs, regardless of whether or not they were possibly related to study drug, is located in the Reported Adverse Event section.
Time Frame: From baseline up to 8 weeks post dose
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo IV | Placebo SC | 0.1 mg LY3016859 IV | 1 mg LY3016859 IV | 10 mg LY3016859 IV | 50 mg LY3016859 IV | 250 mg LY3016859 IV | 750 mg LY3016859 IV | 50 mg LY3016859 SC
Number analyzed (Participants) | 12 | 2 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants
  TEAE | 2 | 0 | 2 | 3 | 0 | 0 | 0 | 1 | 0
  SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacodynamics: Area Under the Concentration-Time Curve (AUC) of Serum Transforming Growth Factor Alpha (TGFα)
Time Frame: Predose up to 8 weeks post dose
Population: All randomized participants who received at least one dose of study drug and had TGFα measurements.
Measure: Mean (Standard Deviation); unit: hour*nanograms/milliliter (h*ng/mL)
Arm/Group | Placebo IV | Placebo SC | 0.1 mg LY3016859 IV | 1 mg LY3016859 IV | 10 mg LY3016859 IV | 50 mg LY3016859 IV | 250 mg LY3016859 IV | 750 mg LY3016859 IV | 50 mg LY3016859 SC
Number analyzed (Participants) | 12 | 2 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hour*nanograms/milliliter (h*ng/mL) | 41271 (109300.8) | 8573 (5072.1) | 2515 (2340.0) | 4444 (4234.6) | 9718 (9089.5) | 4286 (2578.9) | 8244 (6487.5) | 12075 (17137.0) | 10305 (7555.2)

3. Secondary Outcome: Pharmacodynamics: Area Under the Concentration-Time Curve (AUC) of Serum Epiregulin
Time Frame: Predose up to 8 weeks post dose
Population: All randomized participants who received at least one dose of study drug and had serum epiregulin measurements.
Measure: Mean (Standard Deviation); unit: hour*picograms/milliliter (h*pg/mL)
Arm/Group | Placebo IV | Placebo SC | 0.1 mg LY3016859 IV | 1 mg LY3016859 IV | 10 mg LY3016859 IV | 50 mg LY3016859 IV | 250 mg LY3016859 IV | 750 mg LY3016859 IV | 50 mg LY3016859 SC
Number analyzed (Participants) | 12 | 2 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hour*picograms/milliliter (h*pg/mL) | 349927 (118584.0) | 331408 (52233.4) | 280500 (65395.6) | 296022 (94056.4) | 405745 (76219.5) | 379401 (59460.6) | 697442 (229112.6) | 2254733 (1035876.0) | 474081 (280526.0)

4. Secondary Outcome: Pharmacokinetics: Maximum Serum Concentration (Cmax) of LY3016859
Time Frame: Predose up to 8 weeks post dose
Population: All randomized participants who received at least one dose of study drug and had sufficient LY3016859 pharmacokinetic data to estimate Cmax.
Measure: Mean (Standard Deviation); unit: nanograms/milliliter (ng/mL)
Groups:
- 0.1 mg LY3016859 IV: 0.1 milligram (mg) LY3016859 administered once intravenously (IV).
- 50 mg LY3016859 SC: 50 mg LY3016859 administered once subcutaneously (SC).
Arm/Group | 0.1 mg LY3016859 IV | 1 mg LY3016859 IV | 10 mg LY3016859 IV | 50 mg LY3016859 IV | 250 mg LY3016859 IV | 750 mg LY3016859 IV | 50 mg LY3016859 SC
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 6
nanograms/milliliter (ng/mL) | 36 (4.3) | 399 (95.6) | 3812 (718.3) | 18467 (1882.2) | 106967 (20038.0) | 271167 (59650.4) | 3748 (1550.8)

5. Secondary Outcome: Pharmacokinetics: Area Under the Serum Concentration-Time Curve (AUC) of LY3016859 From Time Zero to Infinity (AUC0-inf)
Time Frame: Predose up to 8 weeks post dose
Population: All randomized participants who received at least one dose of study drug and had sufficient LY3016859 pharmacokinetic data to calculate AUC0-inf.
Measure: Mean (Standard Deviation); unit: hour*nanograms/milliliter (h*ng/mL)
Arm/Group | 0.1 mg LY3016859 IV | 1 mg LY3016859 IV | 10 mg LY3016859 IV | 50 mg LY3016859 IV | 250 mg LY3016859 IV | 750 mg LY3016859 IV | 50 mg LY3016859 SC
Number analyzed (Participants) | 0 | 3 | 6 | 6 | 6 | 5 | 5
hour*nanograms/milliliter (h*ng/mL) |  | 9967 (2375.4) | 235759 (46760.1) | 2769626 (516303.9) | 23180633 (9009921.3) | 81450520 (20101546.7) | 1054034 (536160.4)

ADVERSE EVENTS:
Arm/Group | Placebo IV | Placebo SC | 0.1 mg LY3016859 IV | 1 mg LY3016859 IV | 10 mg LY3016859 IV | 50 mg LY3016859 IV | 250 mg LY3016859 IV | 750 mg LY3016859 IV | 50 mg LY3016859 SC
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/2 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/12 | 1/2 | 4/6 | 3/6 | 2/6 | 2/6 | 4/6 | 3/6 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo IV (N=12) | Placebo SC (N=2) | 0.1 mg LY3016859 IV (N=6) | 1 mg LY3016859 IV (N=6) | 10 mg LY3016859 IV (N=6) | 50 mg LY3016859 IV (N=6) | 250 mg LY3016859 IV (N=6) | 750 mg LY3016859 IV (N=6) | 50 mg LY3016859 SC (N=6)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heat rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days